CLINICAL TRIAL: NCT00725322
Title: Subcutaneous Botulinum Toxin for Cutaneous Allodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Assistant Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SU-01072008-965; 11830
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A

ARMS (2):
- Placebo then Botox (Experimental)
  Interventions: Drug: Placebo - Saline
- Botox then Placebo (Experimental)
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Drug: Botulinum Toxin A — Subcutaneous injection of Botulinum Toxin Type A into the patient's scar tissue
  Arms: Botox then Placebo
Drug: Placebo - Saline — Subcutaneous Saline injection given at site of scar neuroma
  Arms: Placebo then Botox

SUMMARY:
Superficial injection of Botulinum toxin has been advocated for cosmetic purposes but has also been reported to be helpful for some pain conditions. The investigators have observed prolonged profound analgesia following subcutaneous superficial injection of Botulinum Toxin Type A (BTA) in patients with certain types of neuropathic pain. The investigators propose to study if addition of BTA extends pain relief compared to placebo when injected subcutaneously into areas of cutaneous allodynia (the property that a normally non-noxious stimulus is perceived as painful).

DETAILED DESCRIPTION:
Post-surgical neuromatous pain patients have marked cutaneous allodynia. Touching their skin with normally non-painful stimuli results in pain. Injected local anesthetics are often effective in providing temporary relief. In the course of clinical practice the investigators have observed that a number of patients with cutaneous allodynia have had marked persistent benefit from subcutaneous injection of Botulinum toxin Type A.

Rather than killing targeted neurons, Botulinum toxin type A inhibits release of acetylcholine from cholinergic nerve terminals in a prolonged but ultimately reversible manner. Neuropathic pain and its hallmark allodynia are classically difficult to treat. Standard treatment with tricyclic antidepressants, anti-epileptic drugs, opiates and spinal cord stimulation is frequently disappointing leaving patients with refractory pain. Surgical or percutaneous ablation of involved nerves has fallen out of favor among many due to disappointing results.

A pilot study is needed to assess the efficacy of superficially injected Botulinum Toxin type A for treatment of cutaneous allodynia and spontaneous pain among patients with neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:- Moderate to severe pain (greater than 4/10) of duration more than 6 months despite previous therapy.

* The patient exhibits at least 80% pain relief following injection of local anesthetic subcutaneously into scar as assessed by change in NRS
* The patient reports the presence of hyperalgesia, allodynia, dysesthesia, or hypoesthesia surrounding the scar
* Age 18-100
* Ability to read, write, and converse in English, provide informed consent, and follow study procedures

Exclusion Criteria:

1. Any neuromuscular disorder such as myasthenia gravis, eaton lambert, muscular dystrophy
2. Any ongoing legal action related to their pain
3. Allergy to local anesthetics
4. A current or history of any severe psychiatric disorder
5. History of any adverse reaction to botulinum toxin
6. History of botulism
7. Untreated infection
8. Coagulopathy
9. Females - positive pregnancy test
10. Surgery within the past 6 months at the site of the painful scar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Carroll, Principal Investigator — Stanford University; Sean Mackey, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 84 total participants were enrolled. 46 were withdrawn before randomization due to failure at screening or following protocol. A total of 38 participants were randomized. A total of 30 participants remained for the first injection after 8 were withdrawn due to medication, surgery, or patient decision. A total of 27 participants completed the study.
Groups:
- Placebo Then Botox: Placebo - Saline:
  Subcutaneous Saline injection given at site of scar neuroma
  Botulinum Toxin A:
  Subcutaneous injection of Botulinum Toxin Type A into the patient's scar tissue Both scar neuroma and scar tissue are locations of cutaneous allodynia in participants. In other words, both injections were in areas where the participant already had pain. Both injections were subcutaneous, right under the skin.
- Botox Then Placebo: Botulinum Toxin A:
  Subcutaneous injection of Botulinum Toxin Type A into the patient's scar tissue
  Placebo - Saline:
  Subcutaneous Saline injection given at site of scar neuroma Both scar neuroma and scar tissue are locations of cutaneous allodynia in participants. In other words, both injections were in areas where the participant already had pain. Both injections were subcutaneous, right under the skin.
Period: First Injection Visit
Arm/Group | Placebo Then Botox | Botox Then Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout (28 Days)
Arm/Group | Placebo Then Botox | Botox Then Placebo
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 1
Period: Second Injection Visit
Arm/Group | Placebo Then Botox | Botox Then Placebo
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Botox: Placebo - Saline:
  Subcutaneous Saline injection given at site of scar neuroma
  Botulinum Toxin A:
  Subcutaneous injection of Botulinum Toxin Type A into the patient's scar tissue
- Botox Then Placebo: Botulinum Toxin A:
  Subcutaneous injection of Botulinum Toxin Type A into the patient's scar tissue
  Placebo - Saline:
  Subcutaneous Saline injection given at site of scar neuroma
- Total: Total of all reporting groups
Arm/Group | Placebo Then Botox | Botox Then Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.62 (14.87) | 50.14 (12.48) | 48.44 (13.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time Until Analgesic Failure
Description: Participants made daily NRS reports via Palm Pilot, and "failure" was defined as (Pre-injection baseline NRS) - (Mean NRS for any 3 preceding days) ≤ 0; or 9 months
Time Frame: Each participant was assessed for up to 224 days per intervention (injection) or until they returned to NRS baseline
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Placebo: Placebo - Saline: Subcutaneous Saline injection given at site of scar neuroma
- Botox: Botulinum Toxin A: Subcutaneous injection of Botulinum Toxin Type A into the patient's scar tissue
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 27 | 27
Days | 76.3 (86.82) | 79 (92.12)

2. Secondary Outcome: NRS Score Three Weeks After Injection
Description: The NRS scores range from 0-100, where 0 indicated no pain and 100 indicated the worst pain.
Time Frame: Three weeks after injection
Population: Although 27 participants completed the study, 3 participants were excluded from analysis of the NRS score because they had missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 24 | 24
Units on a scale | 35.5 (20.07) | 34.7 (23.38)

ADVERSE EVENTS:
Description: Adverse Events were not collected in a way that allows for separation by intervention, thus Adverse Events are reported based on the participant's initial group randomization.
Groups:
- Botox Then Placebo: Placebo - Saline:
  Subcutaneous Saline injection given at site of scar neuroma
  Botulinum Toxin A:
  Subcutaneous injection of Botulinum Toxin Type A into the patient's scar tissue Both scar neuroma and scar tissue are locations of cutaneous allodynia in participants. In other words, both injections were in areas where the participant already had pain. Both injections were subcutaneous, right under the skin.
Arm/Group | Placebo Then Botox | Botox Then Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 8/13 | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Then Botox (N=13) | Botox Then Placebo (N=14)
Dry mouth (General disorders) | 3 | 1
Dyspepsia (General disorders) | 2 | 2
Injection site pain (General disorders) | 3 | 9
Headache (General disorders) | 5 | 4
Nausea (General disorders) | 2 | 1
Flu symptoms (General disorders) | 1 | 3
Torticollis (General disorders) | 1 | 0
Arthralgia (General disorders) | 4 | 5
Back pain (General disorders) | 3 | 5
Increased cough (General disorders) | 1 | 2
Increased weakness (General disorders) | 3 | 3
Dizziness (General disorders) | 2 | 3
Rhinitis (General disorders) | 2 | 2
Other (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes